CLINICAL TRIAL: NCT06375395
Title: Research on Improving the Intervention Effect of Negative Memory Through tACS Enhanced Memory Technology
Brief Title: Boosting The Intervention Effect of Negative Memory Through tACS Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Beijing Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Memory Updating Tasks
Record Dates: First submitted 2024-01-01; First posted 2024-04-19 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2023-11

CONDITIONS: Seizures
Keywords: seizure; transcranial alternating current stimulation; neuromodulation; negative memory; neural mechanisms; retrieval practice; working memory
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tACS (Experimental): Those who participate in the treatment group will receive tACS, which lasts for 40 minutes per day on 3 consecutive days.
  Interventions: Device: Active tACS Device
- Sham tACS (Placebo Comparator): Those who participate in the control group will receive sham tACS, which lasts for 40 minutes per day on 3 consecutive days.
  Interventions: Device: Sham tACS Device

INTERVENTIONS:
Device: Active tACS Device — Transcranial Alternating Current Stimulation
  Arms: Active tACS
Device: Sham tACS Device — Placebo Device that simulates active tACS treatment
  Arms: Sham tACS

SUMMARY:
The objectives of this study include: 1) investigating the impact of negative memory substitution on an individual's other intellectual memories (i.e., neutral memories) and the underlying neurocognitive mechanisms; 2) investigating the memory enhancement effect resulting from retrieval practice associated with memory substitution intervention along with an examination of the neurocognitive mechanisms responsible for this enhancement.

DETAILED DESCRIPTION:
This study will adopt two memory updating strategies: retrieval practice and reactivation.

A 5-day memory updating experimental paradigm is used.

1. On the first day, the old memory A-B linkage is learned, where A represents a neutral word and B is either neutral or negative pictures (half of each, randomly scrambled).
2. On the second day, the old memory A-B association is consolidated again, and after a 15-minute break, the new memory A-C association is learned, where A is still the word A used in the old memory A-B association on the first day, and C is the new neutral and negative pictures (half of each, randomly scrambled, and with inconsistent categories of C and B in each pair of AC and AB). Immediately following this, the new memories of the A-C conjunctions are updated using both Retrieval practice and Restudy (control condition) memory strategies.
3. A-C is extracted/learned using both Retrieval practice and Restudy memory strategies on both day 3 and day 4.
4. On the fifth day, memory tests for associative memory strength, gist and detail memory, as well as emotional valence and strength are performed.

ELIGIBILITY:
Eligibility

Inclusion Criteria:

1. 14-60 years old, male or female, Han Chinese;
2. Drug-resistant epilepsy;
3. Required surgical implantation of SEEG electrodes.

Exclusion Criteria:

1. Progressive encephalopathy or progressive structural damage in the central nervous system;
2. Significant heart, liver, renal insufficiency, and other medical diseases;
3. Severe side effects from taking antiepileptic drugs at the time of enrollment and not inappropriate for SEEG;
4. Significant intellectual disability;
5. A history of alcohol and drug abuse;
6. Any contraindication to MRI.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Negative memory retention | Day 5
  The intervention could disrupt retention of associative negative memory and degree of detail of the negative memories in last A-C paired associate memory test.

SECONDARY OUTCOMES:
The negative emotional intensity of negative memory | Day 5
  The negative memories emotional relief as assesses by the Self-Assessment Manikin (SAM) Measure Scales in last A-C paired associate memory test.
  This measure is constant retrieval practice of neutral memories (A-Cneu) will result in negative memories emotional relief (A-Bneg) compared to the restudy condition.
The retention of associated neutral memories as assesses by the proportions of responses of correctly choosing picture category of B picture (A-Bneu) in last A-B paired associate memory test | Day 5
  This measure is continuous rumination of negative memories (A-Cneg) will increase the strength of associated memories (A-Bneu).
The negative emotional intensity of neutral memory | Day 5
  The emotion-diffusing effects of negative memory rumination as assesses by negative emotional intensity of neutral memories (A-Bneu),which is meature by the Self-Assessment Manikin (SAM) Measure Scales. The negative emotional intensity of neutral memories are more negative with constant retrieval practice of negative memories (A-Cneg) that is the emotion-diffusing effects of negative memory rumination.

CONTACTS AND LOCATIONS:
Overall Officials: Guoguang Zhao, Study Director — Xuanwu Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No